CLINICAL TRIAL: NCT00747279
Title: Comparison of Two Strategies for Glycemic Control in Acute Ischemic Stroke
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sao Domingos (Other)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: HSD001
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Carbohydrate restrictive strategy
  Interventions: Other: Carbohydrate restrictive strategy
- 2 (Active Comparator): Intensive insulin therapy
  Interventions: Drug: Intensive insulin therapy

INTERVENTIONS:
Other: Carbohydrate restrictive strategy — Patients will receive intravenous hydration with a glucose free solution (Ringer III) and enteral nutritional formula containing 33.3% carbohydrates, 16.7% proteins and 50% lipids. These patients will receive regular insulin subcutaneously four times daily, aiming to maintain blood glucose levels at least below 180 mg/dl, and in stable patients, ideally below 150 mg/dl.
  Arms: 1
Drug: Intensive insulin therapy — Continuous intravenous regular insulin infusion will be adjusted to maintain glycemic levels at least below 150 mg/dl, and, in stable patients and ideally, between 80 and 120 mg/dl. Patients will be submitted to capillary glycemic measurements every 2 hours. The insulin dose is adjusted according to an algorithm run by nurses and overseen by physicians. These patients will receive glucosaline (5% glucose + 0.9 NaCl) hydration and enteral nutrition with a formula containing 45% carbohydrates, 17% proteins and 38% lipids.
  Arms: 2

SUMMARY:
The purpose of this prospective randomized controlled trial was to compare intensive insulin therapy with a carbohydrate restrictive strategy in patients with acute ischemic stroke evaluating the outcome through the Glasgow Outcome Scale Extended, hospital mortality and NIHSS during the ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with acute ischemic stroke defined as: Abrupt onset of focal neurologic deficit
* No evidence of intracranial hemorrhage at non-contrasted CT scan.

Exclusion Criteria:

* Age below 18
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2007-06

PRIMARY OUTCOMES:
Neurological outcome through the Glasgow Outcome Scale Extended | At least 4 months after hospital discharge

SECONDARY OUTCOMES:
NIHSS during ICU stay | ICU stay
Hospital mortality | Hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil